CLINICAL TRIAL: NCT00795015
Title: Comparison of the Leuven Protocol With the Glucommander for Postoperative Control of Blood Glucose With an Intravenous Insulin Infusion
Brief Title: Comparison of the Leuven Protocol With the Glucommander for Postoperative Control of Blood Glucose With IV Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: David Baldwin MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06010501
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes
Keywords: postoperative blood glucose control; IV insulin infusion
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- leuven (Active Comparator): these patients had their IV insulin controlled by using the protocol adapted from van den Berghe et al. University of Leuven, Belgium, NEJM Nov. 2001
  Interventions: Drug: insulin regular IV infusion; Drug: IV insulin infusion
- glucommander (Active Comparator): these subjects had IV insulin controlled by a computer program called the glucommander described by Davidson, P et al Diabetes Care Oct. 2005
  Interventions: Drug: insulin regular IV infusion; Drug: IV insulin infusion

INTERVENTIONS:
Drug: insulin regular IV infusion — IV insulin was administered by continuous infusion and the rate changed every hour according to the blood glucose level as determined by each of the protocols being compared
Drug: IV insulin infusion — IV insulin was administered by continuous infusion and the rate changed every hour according to the blood glucose level as determined by each of the protocols being compared

SUMMARY:
The investigators are testing whether a written protocol or a computerized program can more effectively control blood glucose after surgery.

DETAILED DESCRIPTION:
In 2002 we adapted the protocol described by Van den Berghe et al. for use in our own surgical intensive care unit (SICU) with a target blood glucose range from 80 to 120mg/dL. After five years of implementation, we were able to achieve a mean BG of 117 mg/dL in the SICU. 2% of glucose values were <60 mg/dL in the SICU. Given the concern of safety while optimizing glycemic control, we investigated the etiologies for these hypoglycemic episodes and have found two frequent risk factors; the failure to consistently measure blood glucose every hour and in patients with end stage renal failure.

We will investigate whether a computer-based algorithm for the titration of IV insulin will translate to better clinical outcomes and less hypoglycemia. Therefore, we will conduct a prospective randomized trial comparing the Glucommander, a computer-based algorithm with our Van den Berghe protocol for titration of IV insulin in patients after cardiovascular or transplant surgery. This computer based algorithm was invented in 1984 in Atlanta by Dr. Davidson and Dr. Steed who have used it in a variety of applications of IV insulin.

ELIGIBILITY:
Inclusion Criteria:

* s/p open heart or kidney or liver transplant surgery

Exclusion Criteria:

* admission blood glucose less than 120 mg/dl

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Percent of blood glucose values in the target range 80-120 mg/dl | first 200 hours post-op in the ICU

SECONDARY OUTCOMES:
Percent of patient days with a low blood glucose, defines as less than 60 mg/dl | 200 hours while in ICU

CONTACTS AND LOCATIONS:
Overall Officials: David Baldwin, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States